CLINICAL TRIAL: NCT05425693
Title: Comparison of the Effects of Three Warm-up Interventions at the Workplace on Pain, Heart Rate, Work Performance and Physical Capacities Among Vineyard Workers - a Protocol Study
Brief Title: Effects of Three Warm-up Interventions at the Workplace Among Vineyard Workers - a Protocol Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Opti'Mouv (Industry)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00012476-2021-06-12-137
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Pain; Injuries
Keywords: Pain / injuries / warm-up intervention / vineyard workers / physical activity
MeSH Terms: conditions — Pain; Wounds and Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: A cluster randomized study will be implemented among French vineyard workers. Four groups of 30 participants will be constituted; corresponding to four different conditions: (1) hybrid warm-up intervention (HWU); (2) dynamic warm-up intervention (DWU); (3) stretching warm-up intervention (SWU); (4) no warm-up intervention (NWU). A total of 120 vineyard-workers will be recruited to participate in the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hybrid warm-up intervention (Experimental)
  Interventions: Other: Hybrid Warm-up
- Dynamic warm-up intervention (Experimental)
  Interventions: Other: Dynamic Warm-up
- Stretching warm-up intervention (Experimental)
  Interventions: Other: Stretching Warm-up
- No warm-up intervention (No Intervention)

INTERVENTIONS:
Other: Hybrid Warm-up — Dynamic + stretching exercises
  Arms: Hybrid warm-up intervention
Other: Dynamic Warm-up — Dynamic exercises
  Arms: Dynamic warm-up intervention
Other: Stretching Warm-up — Stretching exercises
  Arms: Stretching warm-up intervention

SUMMARY:
Background:

Physical activity programs at the workplace have shown positive results on physical capacities and pain for several years. Due to the duration of the training session, the need of instructor, and the need of a place to practice, these programs are commonly complex to implement. For this reason, many of companies, especially companies in manual sectors are turning to another solution, i.e warm-up intervention before work shift. These interventions present on paper numerous advantages such as short duration, no need to specifically allocate a place in companies and the possibility to perform exercises in working clothes… Surprisingly, while positive effects of warm-up interventions on pain, performance physical and psychological capacities, are expansively reported in sport context, effects of workplace warm-up intervention are lacking. Therefore, the aims of this study are (1) to implement such intervention among vineyard-workers, workers highly exposed to heavy physical workload and pain and (2) to assess their effects on physical (pain, strength, flexibility) and psychological (workload) functions and also on work-related outcomes (work performance, readiness to work)

Methods:

A cluster randomized study will be implemented among French vineyard workers. Four groups of 30 participants will be constituted; corresponding to four different conditions: (1) hybrid warm-up intervention (HWU); (2) dynamic warm-up intervention (DWU); (3) stretching warm-up intervention (SWU); (4) no warm-up intervention (NWU). A total of 120 vineyard-workers will be recruited to participate in the study.

Discussion:

The results will provide more evidence about the short-term effects of warm-up interventions at the workplace, and will provide more evidence on which warm-up modality is the most effective on pain, performance, physical and psychological capacities among vineyard workers.

ELIGIBILITY:
Inclusion Criteria:

* working full time
* having at least 1 year of employment in the company

Exclusion Criteria:

- not to present previous surgery in the low back region in the last 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Perceived pain intensity | Pain intensity will be rated for the last 3 months
  Participants will be asked to rate their pain intensity over 15 anatomical locations using a 0-10 numerical rating scale (NRS), where 0 is used to indicate "no pain" while 10 indicate the "worst possible pain".
Perceived pain intensity | Pain intensity will be rated before the warm-up intervention (Time 0)
  Participants will be asked to rate their pain intensity over 15 anatomical locations using a 0-10 numerical rating scale (NRS), where 0 is used to indicate "no pain" while 10 indicate the "worst possible pain".
Perceived pain intensity | Pain intensity will be rated after the warm-up intervention (Time 1)
  Participants will be asked to rate their pain intensity over 15 anatomical locations using a 0-10 numerical rating scale (NRS), where 0 is used to indicate "no pain" while 10 indicate the "worst possible pain".
Perceived pain intensity | Pain intensity will be rated at the beginning of the working activity (Time 2)
  Participants will be asked to rate their pain intensity over 15 anatomical locations using a 0-10 numerical rating scale (NRS), where 0 is used to indicate "no pain" while 10 indicate the "worst possible pain".
Perceived pain intensity | Pain intensity will be rated after the first hour of work (Time 3)
  Participants will be asked to rate their pain intensity over 15 anatomical locations using a 0-10 numerical rating scale (NRS), where 0 is used to indicate "no pain" while 10 indicate the "worst possible pain".
Perceived pain intensity | Pain intensity will be rated after the second hour of work (Time 4)
  Participants will be asked to rate their pain intensity over 15 anatomical locations using a 0-10 numerical rating scale (NRS), where 0 is used to indicate "no pain" while 10 indicate the "worst possible pain".
Perceived pain intensity | Pain intensity will be rated after three hour of work (Time 5)
  Participants will be asked to rate their pain intensity over 15 anatomical locations using a 0-10 numerical rating scale (NRS), where 0 is used to indicate "no pain" while 10 indicate the "worst possible pain".
Work performance | After one hour of work (Time 3)
  number of grapevine pruned
Work performance | After two hours of work (Time 4)
  number of grapevine pruned
Work performance | After three hours of work (Time 5)
  number of grapevine pruned

SECONDARY OUTCOMES:
Handgrip Strength | Before the warm-up intervention (Time 0)
  Handgrip Strength
Handgrip Strength | After the warm-up intervention (Time 1)
  Handgrip Strength
Handgrip Strength | After three hour of work (Time 5)
  Handgrip Strength
Flexibility | Before the warm-up intervention (Time 0)
  Flexibility of the trunk and the hamstrings - Finger to floor test
Flexibility | After the warm-up intervention (Time 1)
  Flexibility of the trunk and the hamstrings - Finger to floor test
Flexibility | After three hour of work (Time 5)
  Flexibility of the trunk and the hamstrings - Finger to floor test
Flexibility | Before the warm-up intervention (Time 0)
  Flexibility of the shoulders - Back scratch test
Flexibility | After the warm-up intervention (Time 1)
  Flexibility of the shoulders - Back scratch test
Flexibility | After three hour of work (Time 5)
  Flexibility of the shoulders - Back scratch test
Heart rate | Time 0
  Heart rate with a heart rate monitor placed on the wrist
Heart rate | Time 1
  Heart rate with a heart rate monitor placed on the wrist
Heart rate | Time 2
  Heart rate with a heart rate monitor placed on the wrist
Heart rate | Time 3
  Heart rate with a heart rate monitor placed on the wrist
Heart rate | Time 4
  Heart rate with a heart rate monitor placed on the wrist
Heart rate | Time 5
  Heart rate with a heart rate monitor placed on the wrist
Readiness to work | Time 1
  Readiness to work was rated subjectively using a 0-10 numerical rating scale, where 0 was used to indicate "not at all ready" and 10 "perfectly ready to work"
Readiness to work | Time 2
  Readiness to work was rated subjectively using a 0-10 numerical rating scale, where 0 was used to indicate "not at all ready" and 10 "perfectly ready to work"
Work quality | Time 5
  Work quality will be assessed by the workers supervisors, with the same 0-10 scale in every company, developed by the research team and a vineyard growing specialist.
Workload | Time 5
  NASA Task Load Index (NASA TLX) is a multi-dimensional scale used to estimate workload from a worker.
Visuomotor reaction time | Time 0
  The FITLIGHT Trainer (FITLIGHT Sports Corp., Ontario, Canada) will be used to measure the visuomotor reaction time (VMRT).
Visuomotor reaction time | Time 1
  The FITLIGHT Trainer (FITLIGHT Sports Corp., Ontario, Canada) will be used to measure the visuomotor reaction time (VMRT).
Visuomotor reaction time | Time 5
  The FITLIGHT Trainer (FITLIGHT Sports Corp., Ontario, Canada) will be used to measure the visuomotor reaction time (VMRT).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Vuillerme, Phd, Study Director — UniversitéGrenobleAlpes
Locations (1):
- OptiMouv, Pauillac, Gironde, France

REFERENCES:
- [Derived] Larinier N, Vuillerme N, Jadaud A, Malherbe S, Giraud E, Balaguier R. Acute Effects of a Warm-Up Intervention on Pain, Productivity, Physical Capacities and Psychological Perceptions Among Vineyard Workers: a Cluster Randomized Trial. J Occup Rehabil. 2024 Mar;34(1):100-115. doi: 10.1007/s10926-023-10134-2. Epub 2023 Aug 28. PMID 37635160